CLINICAL TRIAL: NCT00583583
Title: Emergency/Compassionate Use - AMPLATZER Duct Occluder
Status: No longer available | Type: Expanded Access
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: AGA-004 E/C; G980103
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Patent; Ductus; Arteriosus

INTERVENTIONS:
Device: Device closure with the AMPLATZER Duct Occluder — Device closure with the AMPLATZER Duct Occluder

SUMMARY:
Emergency/compassionate use for the AMPLATZER Duct Occluder

ELIGIBILITY:
Inclusion Criteria:

* Emergency/compassionate use for patients not meeting the inclusion crtieria for the AMPLATZER Duct Occluder clinical trial

Sex: All
Age Groups: Child, Adult, Older Adult